CLINICAL TRIAL: NCT04570683
Title: Laser Immunotherapy With and Without Topical Anti-PD1 in Basal Cell
Brief Title: Laser Immunotherapy With and Without Topical Anti-PD1 in Basal Cell Carcinomas
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Silje Haukali Omland, Principal Investigator, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Eudra-CT: 2019-003310-14
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: BCC - Basal Cell Carcinoma; Immune Response; Immunotherapy; Ablative Fractionated Laser
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AFL monotherapy (Active Comparator): Singe dose AFL as monotherapy, 100 mJ
  Interventions: Device: Ablative fractionated laser
- AFL+nivolumab (Active Comparator): Single dose AFL 100 mJ followed by immediate intratumoral injection of nivolumab 10% 0.1 ml/cm2 tumor
  Interventions: Drug: Nivolumab 10 MG/ML; Device: Ablative fractionated laser
- nivolumab monotherapy (Active Comparator): Intratumoral injection of nivolumab 10% 0.1 ml/cm2 tumor
  Interventions: Drug: Nivolumab 10 MG/ML

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML — Se previously
  Other Names: opdivo
  Arms: AFL+nivolumab; nivolumab monotherapy
Device: Ablative fractionated laser — Se previously
  Arms: AFL monotherapy; AFL+nivolumab

SUMMARY:
The study aim is to assess the immunological and clinical response in basal cell carcinoma (BCC) treated with ablative fractionated laser (AFL) as monotherapy and compare with BCC treated with combination-therapy of AFL and the anti-PD1-drug nivolumab and with nivolumab as monotherapy.

DETAILED DESCRIPTION:
Explorative open label study. Patients and investigators are non-blinded and patients not randomized to interventions.

Three intervention groups:

1. AFL monotherapy (8-10 patients)
2. AFL+intratumoral nivolumab (8-10 patients)
3. Intratumoral nivolumab monotherapy (8-10 patients)

Patients will attend 4 visits Immunological response is determined by immunohistochemistry (IHC) analysis from biopsies taken prior to AFL, AFL+Nivolumab or Nivolumab treatment (baseline) and compared with biopsies 1 week after treatment. Further, comparison of the immunological response of AFL monotherapy with immunological response AFL+Nivolumab and Nivolumab as monotherapy will be performed.

Patients included for AFL as monotherapy will after tumor demarcation receive AFL of the BCC including a 5 mm margin. An occlusive bandage will be applied to the treated area and is to be removed by the patient 24 hours after treatment or after end of secretion/oozing from the treated area.

Patients included for AFL+Nivolumab will after tumor demarcation receive AFL of the BCC including a 5 mm margin, immediately followed by intratumoral injection of Nivolumab. An occlusive bandage will be applied to the treated area and is to be removed by the patient 24 hours after treatment or after end of secretion/oozing form the treated area.

Patients included for monotherapy with Nivolumab will after tumor demarcation get an intratumoral injection of Nivolumab. An occlusive bandage will be applied to the treated area and is to be removed by the patient 24 hours after treatment or after end of secretion from the treated area.

All patients will have a final visit at week 15, around 12 weeks after first treatment, where the clinical response will be evaluated, and treated tumor will be treated following national guidelines for treatment of BCCs.

For subgroups of clinical responders and non-responders tumor will at week 15 be used for multiplex gene expression analysis via nanostring (Pan cancer immune profiling panel).

For all groups, clinical photographs are taken at every study visit. For patients that present with more than one tumor, patients will be invited to participate with all tumors relevant to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Clinical suspicion of BCC or histologically verified BCC at baseline and histologically verified BCC at visit 2, irrespective of histologic subtype with diameter ≥7 mm at baseline.
* Signed informed consent.
* Female subjects of childbearing potential* must be confirmed not pregnant by a negative pregnancy test prior to study treatment and must use a safe contraceptive method

Exclusion Criteria:

* Concomitant treatment with 5-FU or imiquimod
* Concomitant chemotherapeutic treatment
* Concomitant systemic immunotherapeutic treatment, including Prednisolone
* Pregnant or lactating women
* Allergies to anti-PD1
* Patients with a tendency to form keloids
* Other skin diseases or tattoos in the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
immunological response of AFL and nivolumab as monotherapy and AFL+Nivolumab in BCC | 1 week
  IHC as
  * CD8/CD3 ratio
  * CD4+Foxp3+/CD4 ratio
investigate the clinical response of AFL and Nivolumab as monotherapy and AFL+Nivolumab in BCC | 12 weeks
  evaluated by tumor reduction measured in mm and documented by clinical photos

SECONDARY OUTCOMES:
Tolerability of AFL, intratumoral nivolumab and AFL+Nivolumab | 12 weeks
  evaluated as local skin reactions 1 week and 12 weeks after exposure
Detection of intra-tumoral Nivolumab | 1 week
  evaluated by ELISA with anti-anti-PD1
Analysis and quantification of PD-L1 expression (tumor cells and TILs) | 2 weeks
  evaluated by IHC

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided